CLINICAL TRIAL: NCT02671669
Title: Empowering Individuals Post-Cardiopulmonary Outpatient Rehabilitation to Continue to Live a Heart Healthy Lifestyle: Utilizing Mobile Health Technology
Brief Title: Cardiopulmonary Outpatient Rehabilitation Using Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-01809
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Disease; Pulmonary Disease; Cardiopulmonary Disease
MeSH Terms: conditions — Heart Diseases; Lung Diseases; Pulmonary Heart Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (Active Comparator)
  Interventions: Behavioral: Usual Care
- Movn application (MVN) (Active Comparator)
  Interventions: Behavioral: Movn application (MVN)

INTERVENTIONS:
Behavioral: Usual Care — Discharge packet of Heart Healthy instructions, with self-report health status, quality of life and psychosocial questionnaires, as well as other educational handouts, exit interview to review exercise progress, receive referrals to additional medical services they might need after discharge from the program, with physician.
  Arms: Usual Care (UC)
Behavioral: Movn application (MVN) — Intervention participants will receive the same discharge packet as the UC group along with their exit interview and will receive the following:
  * Participant individualized Heart Healthy instructions for post-cardiac rehabilitation will be integrated into the MVN application including daily medication reminders, physical activity prompts, educational materials, and patient-reported outcome assessment of behavior and psychosocial status.
  * Text messages will be used on an ad hoc basis to provide positive feedback to the participant; two-way messaging between the participant and the research coordinator will be available to provide opportunities to answer specific questions.
  Arms: Movn application (MVN)

SUMMARY:
This is a randomized controlled trial of the feasibility and utility of implementing a smartphone application (MVN) to maintain compliance with a Heart Healthy lifestyle after discharge from a cardiac outpatient rehabilitation program. Patients will be randomized into one of two groups: usual care (control: UC) or Movn mobile application (intervention: MVN). This study will improve and strengthen data collection from this at-risk patient population by recording baseline clinical and psycho social measures while gaining insight into self-reporting of physical activity and frequency between the UC and MVN groups.

ELIGIBILITY:
Inclusion Criteria:

* Current participants in The Joan and Joel Smilow Cardiac Rehabilitation and Prevention Center (JJCRPC) of Rusk Rehabilitation Patient within two weeks of completing outpatient cardiac rehabilitation
* Clinically stable: moderate to low risk strata by standardized clinical assessment
* Clinically stable: moderate to low risk strata by standardized clinical assessment
* no infections
* no unstable arrhythmias, aortic stenosis, thrombophlebitis, dissecting aneurysm or symptomatic anemia
* controlled blood pressure-resting diastolic <100 mmHg, systolic <180mmHg
* no uncompensated heart failure NYHA Class 3-4
* stable angina (no chest pain for month)
* no 2nd or 3rd degree heart block
* no uncontrolled high grade exercise induced ventricular ectopy-hemodynamically stable
* Own an iPhone (version 3 or above), an iPad, or an iPod touch (version 4 or higher) or Android phone or tablet
* Ability to use and comfortable with using mobile health technology to monitor physical and psychosocial health
* Is comfortable using mobile applications
* English language fluency
* Ability to provide informed consent

Exclusion Criteria:

* Patients who do not fulfill all inclusion criteria stated above.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in rate of exercise compliance in standard post cardiac rehabilitation compared to the increased rates of exercise compliance observed with the help of smartphone applications | 6 Months
Difference in Diastolic blood pressure in subjects who have received andard post cardiac rehabilitation compared to of exercise compliance observed with the help of smartphone applications | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bushnik, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States